CLINICAL TRIAL: NCT05524324
Title: Cardiac Resynchronization Therapy in Adult Congenital Heart Disease With Systemic Right Ventricle: A Cross-Over Trial
Brief Title: Cardiac Resynchronization Therapy in Adult Congenital Heart Disease With Systemic Right Ventricle: RIGHT-CRT
Acronym: RIGHT-CRT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: APHP211040
Record Dates: First submitted 2022-07-12; First posted 2022-09-01 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Congenital Heart Disease; Systemic Right Ventricle; Congenitally Corrected Transposition of the Great Arteries; Transposition of Great Vessels; Heart Failure Congenital
Keywords: cardiac resynchronization therapy; congenital heart disease; systemic right ventricle; heart failure
MeSH Terms: conditions — Heart Defects, Congenital; Congenitally Corrected Transposition of the Great Arteries; Transposition of Great Vessels; Heart Failure | interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Intervention Model Description: Double blind randomized cross-over trial. Two cross-over periods of 3 months comparing biventricular pacing (CRT ON) vs. inactive pacing (ventricular back-up pacing or left ventricular pacing alone in patients requiring pacing, CRT OFF), each period in random order.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CRT ON (biventricular pacing) / CRT OFF (inactive or univentricular pacing) (Other): Patients with heart failure and SRV and who have a dispositif CRT will be screened for eligibility. If they are eligible and accept to participate (signed informed consent), the order of activation or inactivation of the CRT will be assigned by randomization.Patients randomized into this arm will start the study in "CRT ON" then "CRT OFF" mode.
  Interventions: Device: CRT ON (biventricular pacing) / CRT OFF (inactive or univentricular pacing)
- CRT OFF (inactive or univentricular pacing) / CRT ON (biventricular pacing) (Other): Patients with heart failure and SRV and who have a dispositif CRT will be screened for eligibility. If they are eligible and accept to participate (signed informed consent), the order of activation or inactivation of the CRT will be assigned by randomization.Patients randomized into this arm will start the study in "CRT OFF" then "CRT ON" mode.
  Interventions: Device: CRT OFF (inactive or univentricular pacing) / CRT ON (biventricular pacing)

INTERVENTIONS:
Device: CRT ON (biventricular pacing) / CRT OFF (inactive or univentricular pacing) — Patients randomized to the CRT ON / CRT OFF arm will undergo a first intervention to activate their device and then a second intervention for 3 months to inactivate their device.
  Arms: CRT ON (biventricular pacing) / CRT OFF (inactive or univentricular pacing)
Device: CRT OFF (inactive or univentricular pacing) / CRT ON (biventricular pacing) — Patients randomized to the CRT OFF / CRT ON arm will undergo a first intervention to inactivate their device and then a second intervention for 3 months to activate their device.
  Arms: CRT OFF (inactive or univentricular pacing) / CRT ON (biventricular pacing)

SUMMARY:
The main objective of RIGHT-CRT is to assess the impact/efficacy of CRT on functional capacity in ACHD patients with SRV.

DETAILED DESCRIPTION:
This study will be the first to bring evidence on CRT efficacy in ACHD patients with heart failure and SRV. If results are positives, CRT may improve functional capacities and quality of life of patients and will become an option of choice in this population. If results are negatives, futile CRT implantation may be avoided in this population in particular considering potential adverse effects and CRT-related complications.

Double blind randomized cross-over trial. 40 patients will be enroled. Their follow-up will be 6 months.

ELIGIBILITY:
Inclusion Criteria:

* systemic right ventricle (SRV),
* CRT-P or CRT-D device implanted for at least 1 month,
* Age ≥18 years old,
* One of the two following CRT indications:

  * NYHA II-IV, right ventricular ejection fraction ≤ 35% and spontaneous QRS duration ≥ 150 ms Or
  * NYHAI-IV, atrioventricular conduction disorders with ventricular pacing > 40% (regardless right ventricular ejection fraction).
* Affiliation to a french social security system (beneficiary or legal)
* Informed and signed consent

Exclusion Criteria:

* Pregnancy or breastfeeding
* Women of childbearing potential who do not have a negative pregnancy test and do not use one of the following methods of birth control: hormonal contraception or intrauterine device or bilateral tubal occlusion
* Patient benefiting from a measure of legal protection (guardianship, curatorship, under judicial safeguard, activated future protection mandate and family authorization),
* Cardiac surgery during the last 3 months or planned during the next 6 months,
* Percutaneous structural cardiac intervention planned during the next 6 months,
* Persistent atrial arrhythmia with catheter ablation planned during the next 6 months,
* Acute congestive heart failure,
* Dysfunction of at least one CRT device lead that compromise biventricular pacing,
* Patient on AME
* Current participation in another interventional clinical study or being in the exclusion period at the end of a previous study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
6-minute walk test | Change from the end of the first cross over period (3 months) to the end of the second cross over period (6 months)
  The 6-minute walk test will be performed by a trained technician, indoors, along a long, flat, straight, enclosed corridor with a hard surface and a minimal length of 30 meters. The length of the corridor will be marked every 3 meters and the turnaround points will be marked with a cone. The starting line will be marked on the floor using brightly colored tape. Specific and standardized instructions will be transmitted to the patient.

SECONDARY OUTCOMES:
Peak oxygen uptake | Change from the end of the first cross over period (3 months) to the end of the second cross over period (6 months)
  VO2 max (ml/kg/min) during exercise test with standardized protocol,
NYHA classification | Change from the end of the first cross over period (3 months) to the end of the second cross over period (6 months)
  NYHA classification (class I to IV)
Right ventricular ejection fraction | Change from the end of the first cross over period (3 months) to the end of the second cross over period (6 months)
  Right ventricular ejection fraction assessed by echocardiography (%)
Tricuspid valve regurgitation | Change from the end of the first cross over period (3 months) to the end of the second cross over period (6 months)
  Tricuspid valve regurgitation grade (I to IV) assessed by echocardiography
QRS duration | Change from the end of the first cross over period (3 months) to the end of the second cross over period (6 months)
  QRS duration measured on electrocardiogram
Quality of life of patients | Change from the end of the first cross over period (3 months) to the end of the second cross over period (6 months)
  Minnesota living with heart failure and SF36v2 questionnaires
BNP | Change from the end of the first cross over period (3 months) to the end of the second cross over period (6 months)
  BNP level
Heart failure | Change from the end of the first cross over period (3 months) to the end of the second cross over period (6 months)
  Number of hospitalizations for heart failure
Diuretics | Change from the end of the first cross over period (3 months) to the end of the second cross over period (6 months)
  Dose of diuretics prescribed
Premature cross-over phase termination | Change from the end of the first cross over period (3 months) to the end of the second cross over period (6 months)
  Number of patients with need for premature cross-over phase termination to restore previous pacing settings
Ventricular arrhythmias | Change from the end of the first cross over period (3 months) to the end of the second cross over period (6 months)
  Number of non-sustained and sustained ventricular arrhythmias

CONTACTS AND LOCATIONS:
Overall Officials: Victor WADLMANN, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (13):
- France (13):
  - CHU de Caen, Caen
  - Hôpital Marie-Lannelongue, Le Plessis-Robinson
  - CHU de Lille, Lille
  - Hôpital Louis Pradel, Lyon
  - Hôpital La Timone, Marseille
  - CHU de Montpellier, Montpellier
  - CHU de Nantes, Nantes
  - Ap-Hp Hegp, Paris
  - AP-HP, Pitié-Salpétrière, Paris
  - CHU de Rouen, Rouen
  - CHU de Toulouse, Toulouse
  - Clinique Pasteur, Toulouse
  - CHU de Tours, Tours

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in publication could be shared. IPD detailed in the protocol of a planned metaanalysis could be shared
Supporting Information: Study Protocol
Time Frame: Two years after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on a scientific project and scientific involvement of the PI team. Collaboration will be fostered. Data sharing must respect the agreements made with funders. Teams wishing obtain IPD must meet the sponsor and IP team to present scientific (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractual agreement. Processing of shared data must comply with European General Data Protection Regulation (GDPR).